CLINICAL TRIAL: NCT06041828
Title: Impact of Regular Home-use Dual Light Photodynamic Therapy in the Prevention of Osteolysis After Dental Implant Surgery
Brief Title: Regular Home-use Dual Light Photodynamic Therapy in the Prevention of Osteolysis After Dental Implant Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been temporarily halted due to time constraints at the study site.
Sponsor: Koite Health Oy (Industry)
Collaborators: Hammaslääkärit Eteläranta 10 (Unknown); University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LumOsteo
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Osteolysis; Dental Implants
Keywords: Lumoral; Dental implant; Osteolysis; Anti-bacterial photodynamic therapy; Oral hygiene
MeSH Terms: conditions — Osteolysis

STUDY DESIGN:
Intervention Model Description: Randomized clinical study on a medical device.
Who Masked: Outcomes Assessor
Masking Description: Data will be collected using individual study codes for participants. Study codes do not reveal which group the participant has belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Standard oral hygiene and Lumoral Treatment home-use
  Interventions: Device: Lumoral Treatment; Other: Standard oral hygiene
- Control group (Active Comparator): Standard oral hygiene only
  Interventions: Other: Standard oral hygiene

INTERVENTIONS:
Device: Lumoral Treatment — Photodynamic antibacterial dual-light device with a marker substance
  Arms: Study group
Other: Standard oral hygiene — Standard oral hygiene instructions

SUMMARY:
The aim of the study is to determine whether regular use of the antibacterial, photodynamic, CE-marked Lumoral device reduces the risk of osteolysis after dental implant surgery. The study also aims to find out whether Lumoral treatment can replace the use of chlorhexidine. Subjects will be randomized into two groups (20 + 20 subjects) and all will be given individual guidance on maintaining good oral hygiene. The participants in the study group will also be given Lumoral appliances with instructions for use at home. The Lumoral device has been shown in previous studies to be safe to use and effective in eliminating harmful oral bacteria.

DETAILED DESCRIPTION:
After a dental implant procedure, implant stability is crucial for the success of the implant. The initial stability of the implant is determined by various factors such as implant design, surgical technique, bone quality, and quantity.

During the implant procedure, the implant is placed into the jawbone and is in direct contact with the surrounding bone. Over time, the bone will grow and fuse with the implant surface in a process called osseointegration. The implant stability is evaluated immediately after the surgery by measuring the implant stability quotient (ISQ) using a device called an implant stability meter.

The ISQ value ranges from 0 to 100, with higher values indicating greater implant stability. In general, an ISQ value of 60 or higher is considered to be a good indicator of implant stability. If the initial ISQ value is low, the implant may be at risk of failure due to lack of stability, and additional measures may be necessary to promote osseointegration, such as using bone grafting materials or growth factors.

In the first few weeks after the implant procedure, the implant may experience some initial mobility due to the inflammatory response and remodeling of the bone around the implant. However, with time, the bone will grow and fuse with the implant, providing a stable foundation for dental restoration.

With proper implant placement and regular follow-up care, the incidence of osteolysis can be minimized. Maintaining good oral hygiene practices, such as regular brushing, flossing, and dental check-ups, can help reduce the risk of inflammatory changes around dental implants. In addition, patients are usually advised to avoid placing excessive force on the implant during the healing process to prevent any damage to the implant and to ensure successful osseointegration. For example, patients can be advised to have a soft food diet at least for a few days after the implant placement.

One of the key issues in maintaining good oral health is patient self-management. A new tool "Lumoral Treatment" has been introduced in order to enhance oral home care. The Lumoral Treatment is a CE-marked medical device developed to provide a potent, targeted antibacterial action on the dental plaque in a home environment. It is used together with the mechanical cleaning (such as toothbrushing) of teeth. The device mechanism of action is antibacterial photodynamic therapy (aPDT) and thus non-medicinal. The Lumoral Treatment includes a light-activated Lumorinse mouth rinse and a Lumoral light activator. Its effect is based on a photodynamic method where the light-sensitive substance - indocyanine green - contained in the Lumorinse mouth rinse is attached to the bacterial film (plaque) and is activated by antibacterial dual light with 405 and 810 nanometers (nm).

The 810 nm light can also have a photobiomodulation effect in promoting bone growth and regeneration. Photobiomodulation (PBM) is a non-invasive therapy that uses low-level light therapy (LLLT) to stimulate cellular function and enhance tissue repair. Near-infrared (NIR) light is one of the commonly used wavelengths for PBM due to its ability to penetrate deeper into tissues. In the case of dental bone, PBM with NIR light has shown promising effects in promoting bone growth and regeneration. In dental applications, PBM with NIR light has shown promise in promoting bone growth and regeneration in cases of dental implant placement, tooth extraction, and periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥ 18 years
* Generally healthy,
* At least one new implant inserted
* New implant inserted
* Agreement to participate in the study with a written consent form signed

Exclusion Criteria:

* Uncontrolled diabetes mellitus (DM)
* Active smoking
* Any significant systemic disease
* Immediate implantation after tooth extraction
* Use of antibiotics within 4 weeks week prior study
* Presence of any physical limitation or restriction that might restrict Lumoral use
* Pregnancy or lactation
* History of six months use of antimicrobials, bisphosphonates, or corticosteroids.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of osteolysis around dental implants | 4 months
  Assessing overall number of study subject that have developed osteolysis

SECONDARY OUTCOMES:
Active matrix metalloproteinase 8 (aMMP-8) | 4 months
  Change in periodontal inflammation marker aMMP-8. The aMMP-8 marker analysis will be performed using Periosafe chairside test (Dentognostics GmbH) according to the manufacturer's instructions.
Bleeding on probing (BOP) | 4 months
  Change in bleeding on probing (BOP)
  A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent" BOP is reported as the percentage (%) of sites with positive findings Calculation formula: number of bleeding sites/ 6 times number of teeth
Probing Pocket Depth (PPD) | 4 months
  Change in the Probing Pocket Depth (PPD)
  A full-mouth assessment, measured at 4 sites per tooth Assessed from the base of the pocket to the gingival margin (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Timo Sorsa, Professor, Principal Investigator — University of Helsinki
Locations (1):
- Hammaslääkärit Eteläranta 10, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dompe C, Moncrieff L, Matys J, Grzech-Lesniak K, Kocherova I, Bryja A, Bruska M, Dominiak M, Mozdziak P, Skiba THI, Shibli JA, Angelova Volponi A, Kempisty B, Dyszkiewicz-Konwinska M. Photobiomodulation-Underlying Mechanism and Clinical Applications. J Clin Med. 2020 Jun 3;9(6):1724. doi: 10.3390/jcm9061724. PMID 32503238
- [Background] Gupta R, Gupta N, Weber, DDS KK. Dental Implants. 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470448/ PMID 29262027
- [Background] H H, G W, E H. The clinical significance of implant stability quotient (ISQ) measurements: A literature review. J Oral Biol Craniofac Res. 2020 Oct-Dec;10(4):629-638. doi: 10.1016/j.jobcr.2020.07.004. Epub 2020 Aug 14. PMID 32983857
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Pandey C, Rokaya D, Bhattarai BP. Contemporary Concepts in Osseointegration of Dental Implants: A Review. Biomed Res Int. 2022 Jun 14;2022:6170452. doi: 10.1155/2022/6170452. eCollection 2022. PMID 35747499
- [Background] Swami V, Vijayaraghavan V, Swami V. Current trends to measure implant stability. J Indian Prosthodont Soc. 2016 Apr-Jun;16(2):124-30. doi: 10.4103/0972-4052.176539. PMID 27141160
- [Background] Qu C, Luo F, Hong G, Wan Q. Effects of photobiomodulation therapy on implant stability and postoperative recovery: a systematic review and meta-analysis. Br J Oral Maxillofac Surg. 2022 Jun;60(5):e712-e721. doi: 10.1016/j.bjoms.2022.01.014. Epub 2022 Feb 5. PMID 35490059
- [Background] Wang Y, Zhang Y, Miron RJ. Health, Maintenance, and Recovery of Soft Tissues around Implants. Clin Implant Dent Relat Res. 2016 Jun;18(3):618-34. doi: 10.1111/cid.12343. Epub 2015 Apr 15. PMID 25873299
- See also: Amengual-Peñafiel. Osteoimmunology drives dental implant osseointegration: A new paradigm for implant dentistry. Japanese Dental Science Review 57 (2021) 12-19. — https://doi.org/10.1016/j.jdsr.2021.01.001
- See also: Elias. Factors Affecting the Success of Dental Implants. Implant dentistry, Aug 2011. DOI: 10.5772/18746 — https://doi.org/10.5772/18746
- See also: Gupta et al. Implant Stability Quotient (ISQ): A Reliable Guide for Implant Treatment. Current Concepts in Dental Implantology. 2021. DOI: 10.5772/intechopen.101359 — https://www.intechopen.com/chapters/79724